CLINICAL TRIAL: NCT01243931
Title: Optical Coherence Tomography Guided Transepithelial Phototherapeutic Keratectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, : David Huang, MD, PhD, Professor of Ophthalmology, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB #00006612-PTK; R01EY018184 (NIH)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Corneal Opacity
Keywords: Phototherapeutic keratectomy; Optical coherence tomography; Corneal opacity; Corneal dystrophy
MeSH Terms: conditions — Corneal Opacity; Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): OCT is assisting in surgery guidance.
  Interventions: Drug: OCT-guided laser phototherapeutic keratectomy

INTERVENTIONS:
Drug: OCT-guided laser phototherapeutic keratectomy — Preoperative measurements from the OCT are used to assist the calculation in deciding the laser depth settings for removal of anterior corneal opacities and defects in the phototherapeutic PTK procedure. The surgeon uses the OCT data to plan a range of treatment parameters to remove most of the opacity while preserving at least 250 microns of residual corneal stroma.
  Other Names: Manufacturer/Name OCT Technology 510(K); Optovue/RTVue-CAM Fourier-domain K071250; Bioptigen/Bioptigen Fourier-domain K063343; Zeiss/Visante Time-domain K051789

SUMMARY:
Optical Coherence Tomography (OCT) machines are non-contact instruments that can measure the depth of scars and other causes of cloudiness in the front of the cornea. The purpose of this study is to determine whether OCT-guided settings for the lasers used for removal of corneal scars and other partial-thickness corneal defects result in improved vision in patients receiving these procedures.

DETAILED DESCRIPTION:
The long-term goal of this project is to utilize newly available very high-speed OCT technology to guide surgical treatments of corneas with superficial opacities and irregularities. OCT is well known for its exquisite resolution, but until recently it has not had sufficient speed to capture the shape of the cornea because of eye motion during OCT scanning. The development of Fourier-domain OCT (FD-OCT) technology has made the requisite speed possible.

Eyes with superficial opacities (corneal scars and stromal dystrophies) can be treated by phototherapeutic keratectomy (PTK). Currently, many surgeons rely on subjective slit-lamp impression of opacity depth to guide PTK and repeat slit-lamp examinations during surgery to determine if the opacity has been sufficiently reduced. Unpredictable hyperopic shifts can occur after PTK. The aim of this project is to develop methods for imaging the cornea with an FD-OCT system that will precisely measure corneal shape and use this information to guide surgery. Patients with irregularly shaped corneas could have their vision restored by reshaping the corneas with a procedure that combines the precision of OCT and lasers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vision primarily limited by superficial opacities and irregularities that could be removed by PTK while leaving at least 250 µm.

Exclusion Criteria:

* Inability to give informed consent
* Inability to maintain stable fixation for OCT imaging
* Inability to commit to required visits to complete the study
* Deep corneal opacities and irregularities
* Cataracts, retinal disease, glaucoma, or other eye conditions that may limit the visual outcome after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in best spectacle-corrected visual acuity (BSCVA) after PTK | 12 months post-procedure
  The primary goal of the trial is to determine the efficacy of the OCT-guided PTK treatment of corneal opacities. During the course of the trial, we will compare the predictive accuracy of the original OCT-guided PTK planning system to the OCT topography-guided system. BSCVA will be measured in typical Snellen acuity notation as 20/xx (feet)

SECONDARY OUTCOMES:
Improvement in uncorrected visual acuity (UCVA), refractive error, and higher order aberrations | 12 months post-procedure
  A second goal is to develop a more sophisticated OCT guidance system incorporating OCT topography of anterior and posterior corneal surfaces and to develop a mathematical model that relates epithelial thickness variation to corneal mean curvature. During the course of the trial, we will compare the predictive accuracy of the original OCT-guided PTK planning system to the OCT topography-guided system. UCVA will be measured in typical Snellen acuity notation as 20/xx (feet)

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Casey Eye Institute, Oregon Health & Science University
Locations (1):
- Casey Eye Institute, Oregon Health & Science University, Portland, Oregon, United States